CLINICAL TRIAL: NCT02707835
Title: The Effect of Edema Control in Patients With Cancer-comparison of Manual Lymph Drainage and Epidermis Fascia Taping With Ultrasonography
Brief Title: Edema Control in Patients With Breast Cancer-comparison of Manual Lymph Drainage and Epidermis Fascia Taping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201505100RIND
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: Edema,taping,ultrasound
MeSH Terms: conditions — Breast Neoplasms; Edema | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group (Active Comparator): self massage, skin care education, manual lymph drainage exercise, compression garment
  Interventions: Other: self massage
- manual lymph drainage group (Active Comparator): manual lymph drainage by a physical therapist, skin care education, manual lymph drainage exercise, compression garment
  Interventions: Other: manual lymph drainage
- experimental group (Experimental): epidermis fascia taping by a physical therapist, skin care education, manual lymph drainage exercise, compression garment
  Interventions: Other: epidermis fascia taping

INTERVENTIONS:
Other: self massage — self massage, skin care education, manual lymph drainage exercise, compression garment
  Arms: control group
Other: manual lymph drainage — manual lymph drainage by a physical therapist, skin care education, manual lymph drainage exercise, compression garment
  Arms: manual lymph drainage group
Other: epidermis fascia taping — epidermis fascia taping by a physical therapist, skin care education, manual lymph drainage exercise, compression garment
  Arms: experimental group

SUMMARY:
The ultrasound imaging could be used to examine the thickness of dermis and the space between dermis and subcutaneous tissue. Whether the measurement of ultrasound imaging correlate to other measurement of edema is unknown.

The purpose of this study is to investigate

1. The reliability of measurement of edema using ultrasound imaging, and the correlation of measurement of ultrasound with other measurement tools.
2. The different effect of edema control by manual lymph drainage technique and epidermis taping technique, and the cost-effective assessment.

Our hypothesis :

1. The measurement of edema with ultrasound imaging is a reliable method and correlate with other edema measurement with moderate correlation.
2. Ultrasound measurement could demonstrate different effect of manual lymph drainage and epidermis taping, and different cost-effectiveness analysis.

ELIGIBILITY:
Inclusion criteria:

1. age:20~80 y/o
2. female patients with unilateral breast cancer after surgery
3. unilateral lymph edema ( circumference of affected side 2cm bigger than sound side）
4. do not receive any treatment of lymph edema Exclusion criteria

1. skin problems on affected side 2. neurological sign involved affected side, ex:stroke, brachial plexus impairment 3. involved other diseases may cause extremity edema, ex: heart failure or chronic kidney disease (stage one to stage five) 4. have medicine which may cause extremity edema 5. pregnant

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
thickness of epidermis and dermis | 10 mins

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Lan Yang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan